CLINICAL TRIAL: NCT05346029
Title: Expanding the Therapeutic Landscape of Post-TIPS Hepatic Encephalopathy
Brief Title: Role of Sarcopenia and Nutritional/Physical Therapy Intervention in Post-TIPS Hepatic Encephalopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anna Baiges (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Hospital Universitario Ramon y Cajal (Other); Gregorio Marañón Hospital (Other)
Responsible Party: Sponsor-Investigator, Anna Baiges, Principal Investigator, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI21/00131
Record Dates: First submitted 2022-04-11; First posted 2022-04-26 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Cirrhosis, Liver; Hepatic Encephalopathy; Sarcopenia
Keywords: Transjugular intrahepatic portosystemic shunt (TIPS); sarcopenia; microbioma; physical therapy; nutrition; hepatic encephalopathy
MeSH Terms: conditions — Liver Cirrhosis; Hepatic Encephalopathy; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to standard medical care or to intervention group for the duration of the study
Masking Description: Due to the nature of the intervention (physical therapy and nutritional optimization) there is no masking in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Patients will be followed-up according to standard clinical practices
- Lifestyle intervention (Experimental): Patients will undergo a 12 week lifestyle intervention (physical therapy and nutritional assessment)
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — Resistance training and nutritional counseling
  Arms: Lifestyle intervention

SUMMARY:
The placement of TIPS (transjugular intrahepatic portosystemic shunt) is the most effective strategy to treat complications of portal hypertension. However, the threat of developing post-TIPS complications diminishes its use and applicability. Hepatic encephalopathy (HE) is the most feared and frequent post-TIPS complication, affecting between 25-54% of patients. Available treatments against HE are only partially effective. Therefore, the best existing strategy is to accurately select patients for TIPS excluding those presenting known high risk factors associated to post-TIPS HE. Despite applying this approach, the incidence of post-TIPS HE still remains very high. The investigators hypothesize that a better identification of risk factors for post-TIPS HE, together with the introduction of therapeutic interventions modulating pathophysiological mechanisms involved in post-TIPS HE development - among which sarcopenia stands out- would lead to a reduction in the incidence of HE and, eventually, to an increase in the number of patients benefiting from TIPS.

Thus, our project is aimed at

1. Demonstrate that a 12 weeks lifestyle intervention based on resistance training and nutritional counseling can reduce sarcopenia and, ultimately, post-TIPS HE.
2. To study predictive factors of post-TIPS HE, focusing on the role of factors that have never been evaluated in the setting of TIPS: gut microbiome and cognitive function

DETAILED DESCRIPTION:
1.- To evaluate the impact of a 12 weeks lifestyle intervention aimed to reduce sarcopenia in post-TIPS hepatic encephalopathy development

The first aim of the study will be approached by an open-label multicenter two arms randomized clinical trial, conducted in Hospital Clínic de Barcelona, Hospital Universitario Ramón y Cajal and Hospital Gregorio Marañón.

All cirrhotic patients submitted for elective TIPS in any of these three hospitals will be eligible. Patients fulfilling inclusion criteria and willing to participate will provide written informed consent and will be randomized to intervention or observational group in a 1:1 ratio. The randomization sequence will be generated by computer. The coded treatment assignment will be kept at the coordinating center in sealed, consecutively numbered, opaque envelopes.

All TIPS procedures will be carried out using PFTE-covered stents and using a stepwise dilatation ideally aiming at a final GPP between 10 and 12 mmHg (below 12 mmHg to protect from portal hypertension, over 10 mmHg to avoid post-TIPS HE).

Follow-up visits will be scheduled at 4 weeks, 12 weeks and 6 months post-TIPS. Patients will be followed up until death, liver transplantation or 6 months after TIPS placement.

Primary outcome: development of post-TIPS overt HE within 6 months after TIPS placement. Overt HE will be defined if any grade from 2 to 4 of West Haven Criteria are present: grade 2, fatigue, apathy, flapping tremor, ataxia, slurred speech; grade 3, somnolence, marked disorientation, rigor, stupor; grade 4, coma.

Secondary outcome: 6 months mortality; development of a second episode of overt HE within the first 6 month; development of minimal HE within the first 6 months; time to development of either overt or minimal HE; development of portal complications during follow-up; effects on sarcopenia; need of admission; percentage of follow-up days spent in the hospital.

Sample size The incidence of post-TIPS HE is stablished at 45% . It is assumed that the effects of a lifestyle intervention comprising resistance training and nutritional counseling could achieve a 50% reduction of HE. With a two-sided 5% alpha and power of 80%, a total of 70 study subjects are needed in each group. A total number of 140 patients is a realistic and achievable enrollment in our clinical setting.

Study subjects The study will include patients with clinical, histological or radiological criteria of cirrhosis that need to be treated with an elective TIPS. Exclusion criteria will be pulmonary hypertension, hepatocelular carcinoma out of Milan criteria, severe liver failure or clinical heart failure and impossibility to perform resistance training. Circumstances directly influencing microbiome (use of antibiotics, lactulose, proton pump inhibitors) will be accurately recorded but will not be considered an exclusion criteria in order to truthfully reflect the usual scenario of clinical practice.

Variables to be collected at baseline, 4 weeks and 6 months The tests contained in the protocol are non-invasive. Clinical follow-up does not differ from the usual for any patient undergoing TIPS.

Blood test Fasting venous blood will be analyzed for liver function tests and ammonia, blood count, general biochemistry and coagulation parameters.

Clinical data including cirrhosis etiology, stage of liver disease, renal function and comorbidities.

Sarcopenia assessment: Sarcopenia will be assessed by: measurement of transversal psoas muscle thickness at CT scan, Liver Frailty Index and muscle strength evaluation (maximal isokinetic strength of the knee extensors).

Transversal psoas muscle thickness normalized per height (TPMT, mm/m) will be assessed in CT scans at baseline (taking advantage of CT scan routinely performed before TIPS to evaluate the splanchnic veins and detect possible technical complications) and 6 months post-TIPS. Measurement of transversal psoas muscle thickness has been shown to be an effective tool to objectively evaluate sarcopenia and predict prognosis in cirrhotic patients, with better accuracy than alternatives such as total cross-sectional area of abdominal skeletal muscle and with the clear advantage of being technically easier.

Liver Frailty Index (LFI) Liver Frailty Index has been evaluated in patients with cirrhosis and has been shown to predict mortality in the LT waiting list.

Muscle strength evaluation. Maximal isokinetic strength of the knee extensors will be determined on the non-dominant leg at a velocity of 90º/s. Eight repetitions will be recorded, each test separated by a 15 second rest. The maximal measured torque will be used in all analyses.

Lifestyle Intervention: Resistance training and nutritional counseling vs standard of care (SOC). Data regarding whether patients already perform exercise and which kind, intensity and duration will be collected at baseline through the International Physical Activity Questionnaire. Patients in the intervention group will begin a resistance training program + nutritional counseling. The investigators have set the intervention duration at twelve weeks because it has been proved that a 12 weeks of resistance training increases muscle strength and muscle size in cirrhosis. Sixty minutes sessions (10 minutes of warmup, 40 minutes of limbs and arms strength exercising routine and 10 minutes of cooling down) will be conducted three non-consecutive days per week and will be supervised by a professional physiotherapist. Exercise intensity will be increased and monitored through the Borg subjective Perception of Exertion Scale. The three participating hospitals are referral centers for portal hypertension complications. Some of the patients treated in these hospitals might not live in the same city and might not be able to presentially attend our facilities 3 days per week. To overcome this possible limitation, the physical training plan has been adapted so that two sessions per week will be telematically supervised.

A nutritional status assessment will be carried out, assessing the diagnosis of malnutrition using the GLIM (Global Leadership Initiative on Malnutrition) criteria. The nutritional intervention will be individualized and advised by a dietitian-nutritionist. Nutritional counseling will be aimed at ensuring the required energy and protein intake through dietary enrichment and late evening snacks. In general terms, it will be recommended to aim for an energy intake of 30-35 kcal/kg/day to maintain body weight at times of major stress, and a daily intake of 1.2 - 1.5 g of protein/kg/day to achieve anabolism. Supplementation using a whey protein module will be indicated with the aim to stimulate muscle mass synthesis. Dietary protein intake will be equally distributed in 3 main meals ensuring a minimum of 20-30g protein/meal, and the optimal time for protein supplementation (0.4g/kg) will be indicated after physical training (3 times/week).

Patients included in the SOC will have the same baseline evaluation and follow-up scheduled visits but without performing resistance training and nutritional counseling.

Second aim: identification of more accurate predictive factors of post-TIPS hepatic encephalopathy that will consequently optimize the use of TIPS and open potential future lines of intervention All the baseline data collected for the first aim will be included in the assessment of post-TIPS HE. Furthermore, microbiome analysis and neuropsychological evaluation will be performed.

* Microbiome analysis. Gut microbiome will be analyzed at baseline and 4 weeks post-TIPS. All the samples from the three hospitals will be processed in Hospital Clínic de Barcelona. Fecal samples collection. Fecal samples will be collected following the International Human Microbiome Standards protocol, using when needed an anaerobic generator. Self-collection samples will be preserved in stabilizing solution at room temperature and handed to the biologic laboratory within 24 hours to 7 days after collection. All samples will be homogenized and aliquoted to 200 mg subsamples that will be kept at -80ºC until the analysis. 16sRNA analysis. 16srRNA microbiota analysis will be performed using Multitag sequencing on an Ion Torrent personal genome machine with the objective of determining the microbial taxa that differentiates between patients who develop HE after TIPS placement. Stool DNA will be extracted and will be analyzed using published multitagged pyrosequencing (MTPA) techniques. Microbiota results will be analyzed using Metastats, standard nonparametric tests (Kruskal-Wallis test) and UNIFRAC QIIME (Quantitative Insights Into Microbial Ecology) principle component analyses (PCA) with multiple comparison adjustments. Functionality of microbiota will be assessed using PiCRUST (Phylogenetic Investigation of Communities by Reconstruction of Unobserved States), and results will be compared between groups. Linear discriminant analysis effect size (LEFSe) will be used to determine the taxa that differentiate the groups. Microbial taxa significantly different on LEFSe between the groups will be then introduced into a logistic regression model with clinical variables of defining cognitive impairment. To interrogate the specific taxa at a deeper level, bacterial families that emerge as significant in the prediction of the logistic regression models will be further analyzed at the genus levels to determine the specific genera associated with specific cognitive impairment or with normal cognitive function..
* Neuropsychological function and cognitive reserve will be measured at baseline. At the 4 weeks and 6 months follow-up visit, only neuropsychological function will be assessed.

Tests specifically designed for Minimal HE evaluation: PHES ; EncephalApp Stroop; Critical Flicker frequency threshold; Animal naming test

Other cognitive function tests: Montreal Cognitive Assessment is a screening tool to distinguish patients with mild cognitive impairment from normal population. Digits-span of WAIS-IV evaluates attention and working memory. Vocabulary of WAIS-IV estimates premorbid IQ. Controlled Oral Word Association Test measures verbal fluency and executive function. ROCF assess visuo-constructional abilities and visual memory functions. Rey Auditory Verbal Learning Test evaluates auditory-verbal memory. Wisconsin Card Sorting Test to measure flexibility, categorization and abstract reasoning. Cuestionario Reserva Cognitiva to estimate the CR.

ELIGIBILITY:
Inclusion Criteria:

* All cirrhotic patients submitted for elective TIPS

Exclusion Criteria:

* Contraindication for TIPS placement, contraindication for physical therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of post-TIPS overt HE within 6 months after TIPS placement | 6 months
  Overt HE will be defined if any grade from 2 to 4 of West Haven Criteria are present: grade 2, fatigue, apathy, flapping tremor, ataxia, slurred speech; grade 3, somnolence, marked disorientation, rigor, stupor; grade 4, coma.

SECONDARY OUTCOMES:
6 months mortality; | 6 months
  Death
development of a second episode of overt HE within the first 6 month | 6 months
  Overt Hepatic encefphalopathy
development of minimal HE within the first 6 months | 6 months
  minimal HE detected through PHES neuropsicological test
development of minimal HE within the first 6 months | 6 months
  minimal HE detected through Encephal App Stroop neuropsicological tests
development of minimal HE within the first 6 months | 6 months
  minimal HE detected through Critical Flicker frequency threshold neuropsicological test
development of minimal HE within the first 6 months | 6 months
  minimal HE detected through Animal naming neuropsicological test
time to development of either overt or minimal HE | 6 months
  time to development of either overt or minimal HE
development of portal hypertension complications during follow-up; | 6 months
  ascites, variceal bleeding
effects on sarcopenia | 6 months
  transversal psoas measurement. Measurements will be performed at the level of the umbilicus. Axial psoas muscle thickness and transversal psoas muscle thickness will be measured. All measurements will be performed on the right psoas muscle. Psoas muscle thickness will be normalized by dividing the value by patient's height. Based on data published by Golse et al in 2017, sarcopenia is defined as a TPMT below 1562 mm/m for men and below 1464 mm/m for women
need of admission | 6 months
  hospital admission because of any cause
percentage of follow-up days spent in the hospital | 6 months
  percentage of follow-up days spent in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Anna Baiges, MD, PHD, Principal Investigator — Hospital Clinic of Barcelona
Locations (3):
- Spain (3):
  - Hospital Clínic de Barcelona, Barcelona, Catalonia
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goldbecker A, Weissenborn K, Hamidi Shahrezaei G, Afshar K, Rumke S, Barg-Hock H, Strassburg CP, Hecker H, Tryc AB. Comparison of the most favoured methods for the diagnosis of hepatic encephalopathy in liver transplantation candidates. Gut. 2013 Oct;62(10):1497-504. doi: 10.1136/gutjnl-2012-303262. Epub 2013 Jan 7. PMID 23297006
- [Result] Lauridsen MM, Jepsen P, Vilstrup H. Critical flicker frequency and continuous reaction times for the diagnosis of minimal hepatic encephalopathy: a comparative study of 154 patients with liver disease. Metab Brain Dis. 2011 Jun;26(2):135-9. doi: 10.1007/s11011-011-9242-1. Epub 2011 Apr 12. PMID 21484318
- [Result] Riggio O, Merlli M, Pedretti G, Servi R, Meddi P, Lionetti R, Rossi P, Bezzi M, Salvatori F, Ugolotti U, Fiaccadori F, Capocaccia L. Hepatic encephalopathy after transjugular intrahepatic portosystemic shunt. Incidence and risk factors. Dig Dis Sci. 1996 Mar;41(3):578-84. doi: 10.1007/BF02282344. PMID 8617139
- [Result] Nardelli S, Lattanzi B, Torrisi S, Greco F, Farcomeni A, Gioia S, Merli M, Riggio O. Sarcopenia Is Risk Factor for Development of Hepatic Encephalopathy After Transjugular Intrahepatic Portosystemic Shunt Placement. Clin Gastroenterol Hepatol. 2017 Jun;15(6):934-936. doi: 10.1016/j.cgh.2016.10.028. Epub 2016 Nov 2. PMID 27816756
- [Result] Merli M, Giusto M, Lucidi C, Giannelli V, Pentassuglio I, Di Gregorio V, Lattanzi B, Riggio O. Muscle depletion increases the risk of overt and minimal hepatic encephalopathy: results of a prospective study. Metab Brain Dis. 2013 Jun;28(2):281-4. doi: 10.1007/s11011-012-9365-z. Epub 2012 Dec 7. PMID 23224378
- [Result] Gioia S, Merli M, Nardelli S, Lattanzi B, Pitocchi F, Ridola L, Riggio O. The modification of quantity and quality of muscle mass improves the cognitive impairment after TIPS. Liver Int. 2019 May;39(5):871-877. doi: 10.1111/liv.14050. Epub 2019 Feb 6. PMID 30667572
- [Result] Aamann L, Dam G, Borre M, Drljevic-Nielsen A, Overgaard K, Andersen H, Vilstrup H, Aagaard NK. Resistance Training Increases Muscle Strength and Muscle Size in Patients With Liver Cirrhosis. Clin Gastroenterol Hepatol. 2020 May;18(5):1179-1187.e6. doi: 10.1016/j.cgh.2019.07.058. Epub 2019 Aug 5. PMID 31394282
- [Result] Bajaj JS, Betrapally NS, Gillevet PM. Decompensated cirrhosis and microbiome interpretation. Nature. 2015 Sep 17;525(7569):E1-2. doi: 10.1038/nature14851. No abstract available. PMID 26381988